CLINICAL TRIAL: NCT06403345
Title: A Feasiblity Study of Green Activity Program for People Living With Memory Challenges
Acronym: GAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: American Federation for Aging Research (Other)
Responsible Party: Principal Investigator, Rebecca Lassell, Assistant Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22206
Record Dates: First submitted 2024-04-26; First posted 2024-05-07 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease; Subjective Cognitive Decline (SCD)
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm pre/post study (Experimental): GAP 12-week Intervention for People Living with Memory Loss & Study Partners involves an evaluation, goal-setting, coaching and strategy training over 4-8 virtual or phone sessions for 30-90 minutes each over 12 weeks, with 2 phone or virtual check-ins for 15-30 minutes.
  GAP Intervention Outdoor Activity Professionals involves a site-evaluation (Accessibility, Fall risk) and education on Dementia Training, SMART Goal setting, Strategy Training for Tailoring Nature Activities, and Behavioral Activation strategies with support from the OT.
  Interventions: Behavioral: Green Activity Program

INTERVENTIONS:
Behavioral: Green Activity Program — See arm description.

SUMMARY:
The purpose of this study is to test the Green Activity Program that was designed with people living with memory challenges and their study partners to see if it can be done and if they enjoy the program. "Green activities" are nature activities that the person enjoys and can be done with other people or pets. For example, dog walking, hiking, outdoor yoga, and gardening are all green activities. The purpose of the program is to help people living with memory challenges participate in nature activities they enjoy. The goal of the program is to help people stay active and improve their health and well-being.

DETAILED DESCRIPTION:
This is a single arm pre/post feasibility study lasting up to 1 year. Investigators will recruit in n=40 dyads (people living with memory challenges and their study partners n=80 total) and expect n=30 (n=60 total people living with memory challenges and study partners) to complete the 12-week GAP and evaluate it for feasibility and acceptability. Anonymous program evaluation surveys will be administered either via paper or RedCap survey to the outdoor activity professionals who participated in the study. Brief recorded phone interviews (5 minutes) will be conducted with the people living with memory challenges and their study partners after the intervention and 15-minute brief calls with the outdoor activity professionals will be used to gather feedback to refine the program. Informal conversations with the occupational therapist(s) delivering the intervention will occur to identify areas for refinement and will be documented with anonymous notes and no identifiable data collected from them. Sustained behavior change will be measured in people living with memory challenges at 4 weeks after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 45 years or older
* Has memory challenges or difficulties thinking
* Have access and ability to respond to the telephone (mobile or landline)

Study partner

* 18 years or older
* Speaks Spanish or English
* Identified by the PLMC as a person they feel comfortable with who they would like to join them in the study. The study partner's participation is based on level of support needed for the PLMC.

Outdoor activity professionals

* 18 years or older
* at least 1 year experience providing outdoor activities

Exclusion Criteria:

Participants living with memory challenges will be excluded if they do not meet inclusion criteria or if they indicate any of the following on the 2023 Physical Activity Readiness Questionnaire + (PAR-Q+) :

* Heart failure or, difficulty controlling Coronary Artery Disease, Diagnosed Abnormality of Heart Rhythm, or other cardiovascular condition.

  * If they report difficulty controlling CAD, Diagnosed abnormality of heart rhythm they will be excluded.
  * If they endorse a diagnosis of heart failure, AND report symptoms greater than NYHA Functional Classification Stage I: "No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation or shortness of breath," they will be excluded. Research assistants will be trained to ask about these symptoms during usual activities of daily living.
  * If their doctor has told them not to participate in physical activity due to their heart condition or another medical condition, they will be excluded.
* Cancer and are in an active cycle of infusion chemotherapy or daily radiation treatments.

  * People with cancer whose treatment regimen does not impact their day to day routines (e.g.-oral chemotherapy agents) may participate. Research assistants will be trained to ask about the impact of cancer and cancer care on day to day activities and physical activity.
  * If their doctor has told them not to participate in physical activity due to their cancer or cancer treatment or another medical condition, they will be excluded.
* Experienced a black out, fainted, or lost consciousness as a result of a head injury in the past 12 months.
* Often experienced signs and symptoms of low blood sugar (hypoglycemia) following exercise and/or daily activities.
* 2 or more hospitalizations in 6 months

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility intervention completion rate | Through study completion
  intervention completion rate of 75%
Other Feasibility measures | Through study completion
  75% attendance, 75% retention, intervention fidelity using a checklist by an outside rater with at least 75% of potential active ingredients present in 25% of randomly sampled sessions: tailoring (environment, activity, personalized delivery), behavioral activation, and nature (outdoor environment or incorporating nature [plant or animal]). Feasibility data of recruitment rates (eligible participants/# recruited per month), feasibility of assessments (time to complete, with an 80% completion rate) will be collected, and we will also track missing data.
Acceptability | Up to one month after the 12-week program.
  Two selected questions from the Intervention Tolerability scale will be asked to the person living with memory challenges over the phone: "The program was easy to use" and "I liked this program." Rated by (yes/no). We expect at least 70% of people living with memory challenges will be satisfied with the intervention (yes to both questions).

SECONDARY OUTCOMES:
Goal Attainment Scaling | Up to one month after the 12-week program
  Primary goal met (yes/no)
Quick Physical Activity Scale | Up to 1 month before and after the 12-week program
  Physical activity
Heart Rate | 1 week pre 12-week program and 1 week post
  ActiGraph LEAP
Physical activity | 1 week pre 12-week program and 1 week post
  ActiGraph LEAP
Sedentary time | 1 week pre 12-week program and 1 week post
  ActiGraph LEAP
Health | Up to 1 month before and after the 12-week program
  Patient-Reported Outcomes Measurement Information System: Physical health. Scored on the T-score metric. High scores mean more of the concept being measured.
  A score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population.
Well-being | Up to 1 month before and after the 12-week program
  Patient-Reported Outcomes Measurement Information System: Mental Health. Scored on the T-score metric. High scores mean more of the concept being measured.
  A score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population.
Social Participation | Up to 1 month before and after the 12-week program
  Patient-Reported Outcomes Measurement Information System: Satisfaction with participation in social activities. Scored on the T-score metric. High scores mean more of the concept being measured.
  A score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population.
Depression | Up to 1 month before and after the 12-week program
  Geriatric Depression Scale short form,
Behavioral Activation | Up to 1 month before and after the 12-week program
  Behavioral Activation Scale Short Form
Sleep | 1 week before and 1 week after the 12 week intervention
  ActiGraph LEAP
UCLA 3-item Loneliness scale | Up to 1 month before and after the 12-week program
  Loneliness
Neuropsychiatric symptoms | Up to 1 month before and after the 12-week program
  Neuropsychiatric symptoms questionnaire
Brief phone interviews | Up to 1 month after the 12-week program
  2 -Post questions over the phone: "What did you like about the program? What would you change?"
Study Partner Health | Up to 1 month before and after the 12-week program
  Patient-Reported Outcomes Measurement Information System: Physical health. Scored on the T-score metric. High scores mean more of the concept being measured.
  A score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population.
Study Partner well-being | Up to 1 month before and after the 12-week program
  Patient-Reported Outcomes Measurement Information System: Mental Health. Scored on the T-score metric. High scores mean more of the concept being measured.
  A score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population.
Study Partner Social Participation | Up to 1 month before and after the 12-week program
  Patient-Reported Outcomes Measurement Information System: Satisfaction with participation in social activities. Scored on the T-score metric. High scores mean more of the concept being measured.
  A score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population.
Study Partner Depression | Up to 1 month before and after the 12-week program
  Geriatric Depression Scale short form
Feasibility for Study partner | Up to 1 month after the 12-week program
  Feasibility of an Intervention Measure
Acceptability for Study Partner | Up to 1 month after the program
  Acceptability of an Intervention Measure
Appropriateness for Study Partner | Up to 1 month after the 12-week program
  Appropriateness of an Intervention Measure
Brief phone interview | Up to 1 month after the 12-week program
  "What did you like about the program? What would you change?"
Outdoor Professional Dementia Knowledge | Up to 1 month before and after the dementia training
  Dementia Knowledge Assessment
Outdoor Professional strategies for tailoring activities | Up to 1 month before and after the strategy training
  Strategies for Tailoring Activities quiz
Outdoor Professional brief phone interview | Up to 2 weeks after the 12 week program
  15-minute brief phone interview post
Sustained Behavior Change for People Living with Memory Challenges | 1 month after the 12 week program
  3 Questions asked via phone
  1. Are you still doing the activities?
  2. (If yes) Do you plan to continue doing the activities? (If no) Why not? Do plan to do them in the future?
  3. Have you added any new activities?
Cognitive function | Up to 1 month before and after 12 week program
  T-MoCa
Usability | up to 2 weeks after baseline testing with the ActiGraph LEAP and CenterePointe App software
  Holden's Simplified Systems Usability Scale (SSUS)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Lassell, PhD, Principal Investigator — Indiana Unversity
Locations (1):
- Indiana University Bloomington, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lassell R, Metaxas A, Wang K, Hantgan S, Gottipati P, Zwerling S, Pena T, Pollak C, Gitlin L, Jariwala S. Applying the Human-Centered Innovation Biodesign Framework to the Development and Piloting of a Program to Mitigate Risk for Cognitive Decline Among Historically Underrepresented Individuals: Case Study. JMIR Form Res. 2025 Oct 15;9:e64930. doi: 10.2196/64930. PMID 41092385